CLINICAL TRIAL: NCT03850678
Title: Restoration of Spectral Resolution With Hearing-aid Amplification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 18892; R21DC017588 (NIH)
Record Dates: First submitted 2019-02-18; First posted 2019-02-22 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing Aid (Experimental): Group of participants with hearing loss. Subjects will complete a questionnaire that asks relevant questions about their medical and developmental history and educational level. Participants will be screened for a potential cognitive impairment using the Montreal Cognitive Assessment Basic (MOCA-B). Working memory span will be assessed using the reading span test. Each subject will undergo a routine audiological examination, including audiometric testing and tympanometry. The ability of the subjects to detect different frequencies and to repeat speech presented at a variety of levels, while manipulating different hearing aid parameters and also without the provision of amplification, will be assessed.
  Interventions: Device: Hearing Aid
- Normal Hearing (No Intervention): Group of participants with normal hearing that serve as a reference group. Subjects will complete a questionnaire that asks relevant questions about their medical and developmental history and educational level. Participants will be screened for a potential cognitive impairment using the Montreal Cognitive Assessment Basic (MOCA-B). Working memory span will be assessed using the reading span test. Each subject will undergo a routine audiological examination, including audiometric testing and tympanometry. The ability of the subjects to detect different frequencies and to repeat speech presented at a variety of levels will be assessed.

INTERVENTIONS:
Device: Hearing Aid — Hearing Aid
  Arms: Hearing Aid

SUMMARY:
The objective of this study protocol is to determine the efficacy of using aided measures of spectral resolution to set the dynamic range of hearing with hearing-aid amplification. Measures of spectral resolution will be obtained, as will measures of speech recognition.

DETAILED DESCRIPTION:
Adults with hearing loss are more vulnerable to interference from background noise than adults with normal hearing. Despite the fact that the ability to extract speech information imbedded in background noise requires decoding differences in level across frequency (spectral information), few studies have addressed the extent to which spectral information can be provided to listeners with hearing loss. This fundamental gap in our knowledge prevents society from effectively addressing the systemic effects of hearing loss on communication, income, and ability to socialize with others. This work is a new application of established methods of characterizing spectral resolution to that of the most common device for rehabilitation of hearing loss, hearing-aid amplification. Because hearing aids do not require premarket approval, FDA oversight is not applicable to this clinical trial.

The experiments will examine the degree to which access to spectral information can be restored to adults with hearing loss and the feasibility of utilizing this information to decrease interference from background noise. Aim 1 will delineate the impact of hearing-aid amplification on spectral decoding. Technology options that must be set by the clinician or hearing-aid manufacturer will be examined, including the frequency-specific gain, compressor speed, and number of compression channels. The proposed experiments will test the hypothesis that restoration of the lost dynamic range of hearing can support the encoding of spectral information. It is also hypothesized that the combination of technology options that best restore access to spectral information will differ across individuals and that these differences across individuals can be partially accounted for by an estimate of outer hair cell function. Aim 2 will determine the extent to which restoring access to spectral information supports speech recognition in background noise, under the guiding hypothesis that improving spectral resolution increases speech understanding. If it can be demonstrated that measures of spectral resolution with the provision of amplification are useful at delineating those who stand to benefit from different technology options, the knowledge gained could then be applied to the clinic to allow for clinicians to more successfully choose among different rehabilitation options.

ELIGIBILITY:
Inclusion Criteria:

* normal tympanograms (peak admittance of ≥ 0.2 mmhos, -200 to 50); Hearing thresholds for normal hearing group less than or equal to 20 decibels in hearing level (dB HL) from .25 to 8 kHz. Pure-tone average (2, 4 & 6 kHz) hearing thresholds for participants with hearing loss of 30 - 65 dB HL.

Exclusion Criteria:

* cognitive impairment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Brennan, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- Barkley Memorial Center, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed a questionnaire about their medical and developmental history and educational level. Participants cognitive ability assessed using the Montreal Cognitive Assessment Basic (MOCA-B). Each subject underwent a routine audiological examination, including audiometric testing and tympanometry. Due to not qualifying on basis of inclusion or exclusion criteria (age, degree of hearing loss, or tympanometric findings), 85 participants were excluded before assignment to groups.
Groups:
- Hearing Aid: Group of participants with hearing loss. Working memory span was assessed using the reading span test. The ability of the subjects to detect different frequencies and to repeat speech presented at a variety of levels, while manipulating different hearing aid parameters and also without the provision of amplification, was assessed.
  Hearing Aid: Hearing Aid
- Normal Hearing: Group of participants with normal hearing that serve as a reference group. Working memory span was assessed using the reading span test. The ability of the subjects to detect different frequencies and to repeat speech presented at a variety of levels was assessed.
Period: Overall Study
Arm/Group | Hearing Aid | Normal Hearing
Started | 96 | 28
Completed | 85 | 25
Not Completed | 11 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Experimenter Error | 1 | 1
Not completed — Did Not Condition To Experiment | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Normal Hearing: Group of participants with normal hearing that serve as a reference group.
- Hearing Aid: Group of participants with sensorineural hearing loss who were tested under conditions with hearing aid amplification.
- Total: Total of all reporting groups
Arm/Group | Normal Hearing | Hearing Aid | Total
Number analyzed (Participants) | 25 | 85 | 110
Age, Continuous [Mean (Full Range); unit: years] | 66 [49 to 75] | 70 [43 to 78] | 69 [43 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 47 | 67
  Male | 5 | 38 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 79 | 102
  Unknown or Not Reported | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 23 | 84 | 107
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 25 | 85 | 110
Montreal Cognitive Assessment Basic (MOCA-B) [Mean (Full Range); unit: scores on a scale] — MOCA-B is a measure of cognitive ability that assess aspects of cognitive ability such as executive function, immediate recall, and delayed recall. Each task is scored and then the sum of scores across tasks is computed. The range of possible scores is 0 to 30 (with 30 indicating perfect cognitive ability per this assessment).
  scores on a scale | 26 [23 to 30] | 26 [17 to 30] | 26 [17 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Spectral Resolution
Description: Measure of spectral resolution (Q10) obtained from the fast psychophysical tuning curve test. For this study, Q10 was computed as the target frequency divided by the bandwidth of the tuning curve (10 dB above the threshold at the tip of the tuning curve test). Higher numbers on this scale indicate sharper (better) tuning. The lower limit for this scale is 0 and there is no upper limit.
Time Frame: Each test was approximately 10 minutes and was completed after each experimental manipulation
Population: Consisted of varying conditions and number of participants per condition, including three different compression speeds (instant, fast, slow), three different number of compression channels (4, 8, 16) and two different amplification conditions (unaided, aided).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hearing Aid Group: Participants with hearing loss who were tested with hearing aid amplification.
- Normal Hearing: Comparison group of individuals with normal hearing. This group was only tested without hearing aid amplification (in the unaided condition).
Arm/Group | Hearing Aid Group | Normal Hearing
Number analyzed (Participants) | 68 | 14
units on a scale
  Instant: number analyzed (Participants) | 35 | 0
  Instant | 3.5 (2.2) |
  Fast: number analyzed (Participants) | 35 | 0
  Fast | 3.3 (1.9) |
  Slow: number analyzed (Participants) | 35 | 0
  Slow | 3.2 (1.6) |
  4 Channels: number analyzed (Participants) | 42 | 0
  4 Channels | 2.8 (1.2) |
  8 Channels: number analyzed (Participants) | 42 | 0
  8 Channels | 2.5 (1.7) |
  16 Channels: number analyzed (Participants) | 42 | 0
  16 Channels | 3.5 (1.1) |
  Unaided: number analyzed (Participants) | 14 | 14
  Unaided | 2.7 (1.7) | 3.9 (2.0)
  Aided: number analyzed (Participants) | 14 | 0
  Aided | 3.2 (1.1) |
Statistical Analysis 1: Comparison: Hearing Aid Group; This analysis examined Q10 for those participants who completed the compression speed experiment (instant, fast, slow); Test type: Superiority; p = .774, ANOVA
Statistical Analysis 2: Comparison: Hearing Aid Group; This analysis examined Q10 for those participants who completed the compression channel conditions (4, 8, 16); Test type: Superiority; p < .001, ANOVA
Statistical Analysis 3: Comparison: Hearing Aid Group; This analysis compared Q10 for those participants who completed the unaided and aided conditions; Test type: Superiority; p = .167, ANOVA

2. Primary Outcome: Speech Recognition
Description: measure of spatial release from masking (dB) for a masker presented at 70 dB SPL.
Time Frame: Each test was approximately 10 minutes and was completed after each experimental manipulation
Population: Participants with normal hearing were only tested unaided. Participants with hearing loss were tested unaided, 4 channels with fast compression, and 16 channels with fast compression. Fast compression with 4 and 16 channels were assessed to assess the potential role of changes in spectral resolution to changes in speech recognition between these two conditions.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Normal Hearing | Hearing Aid
Number analyzed (Participants) | 17 | 15
dB
  unaided | 6.6 (5.1) | 4.5 (1.9)
  4 channels: number analyzed (Participants) | 0 | 15
  4 channels |  | 4.0 (3.2)
  16 channels: number analyzed (Participants) | 0 | 15
  16 channels |  | 3.7 (2.8)
Statistical Analysis 1: Comparison: Hearing Aid; Statistical analysis of number of compression channels (unaided, 4 channel, 16 channels); Test type: Superiority; p = .741, ANOVA
Statistical Analysis 2: Comparison: Normal Hearing vs Hearing Aid; Spatial Release from Masking, unaided; Test type: Superiority; p = .062, t-test, 1 sided — Due to Levene's Test for Equality of Variances, equal variances were not assumed

3. Secondary Outcome: Working Memory
Description: Measure of working memory (correctly repeated words from the reading span test). The minimum (poorer) and maximum (better) values are 0 and 57, respectively.
Time Frame: Each test was approximately 30 minutes and was completed only once per subject.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Hearing | Hearing Aid
Number analyzed (Participants) | 14 | 42
score on a scale | 23.6 (6.8) | 20.1 (7.4)
Statistical Analysis 1: Comparison: Hearing Aid; Linear regression of score for the reading span (independent variable) to Q10 (dependent variable, 16 channel compression condition) for the participants who completed the compression channel experiment; Test type: Superiority; p = .805, Regression, Linear

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Groups:
- Normal Hearing: Group of participants with normal hearing that serve as the reference group.
Arm/Group | Hearing Aid | Normal Hearing
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT03850678/Prot_SAP_000.pdf